CLINICAL TRIAL: NCT02169323
Title: Step-down of Inhaled Corticosteroids (ICS) in Non-eosinophilic Asthmatics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Renaud Louis (Other)
Responsible Party: Sponsor-Investigator, Renaud Louis, Head of the Pneumology Department, University of Liege
Organization: University of Liege (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-98; 2014-001316-19 (EudraCT Number)
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Non-eosinophilic Asthma; Inhaled corticosteroids; Step-down
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Step-down (Experimental): Step-down of the inhaled corticosteroid (ICS) dose
  Interventions: Other: Step-down

INTERVENTIONS:
Other: Step-down — Step-down of the inhaled corticosteroid (ICS) dose until discontinuation for 6 months

SUMMARY:
There is growing evidence that non-eosinophilic asthmatics are less sensitive to inhaled corticosteroids (ICS) than eosinophilic asthmatics.

As non-eosinophilic asthmatic patients are treated by ICS according to international guidelines for asthma, the investigators would like to investigate whether stepping-down of ICS in these patients may be safe. Indeed, the investigators can reasonably expect that a progressive cessation of ICS is possible in some of these patients without any clinical worsening.

DETAILED DESCRIPTION:
For patients whose asthma is not controlled at the beginning of the study, a step-up of the treatment is planned to the step 4 of Global Initiative for Asthma (GINA). This step-up will last for 3 months and will permit to ensure that these patients achieve the best possible level of asthma control. A progressive step-down of the inhaled corticosteroids (ICS) will then be achieved.

For patients whose asthma is controlled at the beginning of the study, a progressive step-down of the ICS will be directly achieved.

The progressive step-down of the ICS dose will be undertaken every 3 months according to the dose levels defined by GINA guidelines (from high to low daily dose) until a complete cessation of the ICS for 6 months. Other associated asthma treatment of asthma will be kept unchanged.

At each quarterly visit, a clinical composite outcome will be measured, for each patient. This composite outcome includes the score of asthma control questionnaire (ACQ) and the number of exacerbations. This outcome will determine at each visit if patients continue the study (success criterion) or stop the study (failure criterion). The success criterion is defined in the section "Current Primary Outcome"

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Physician-diagnosed asthma based on the presence of typical symptoms (wheezing, breathlessness, chest tightness, cough)
* Asthma confirmed by:

  * Forced expiratory volume in 1 second (FEV1) increase of at least 12% and 200 mL after inhalation of 400 mcg salbutamol
  * And/or a provocative concentration of methacholine causing a 20% fall in FEV1 (PC20M) less than 16 mg/ml
* Sputum eosinophils rate less than 3%
* Absolute blood eosinophils count less than 400 per mm3
* Treatment with a stable dose of inhaled corticosteroid (ICS) for the previous three months

Exclusion Criteria:

* High risk of asthma-related death, defined by:

  * Near-fatal asthma history, requiring a stay in an intensive care unit
  * Current using or recent discontinuation (four weeks) of oral corticosteroids (OCS)
* Treatment with omalizumab
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-06; Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patients meeting the success criterion at each visit until the end of the study (corresponding to a discontinuation of the treatment by inhaled corticosteroids (ICS) for 6 months) | Up to 12 months to reach a 6 month stop of ICS
  The success criterion is defined at each visit as:
  - An Asthma Control Questionnaire (ACQ) score lower than 1.5 or a variation of the ACQ score from baseline smaller than 0.5
  AND
  - A number of severe exacerbations from the start of the step-down smaller or equal to the number of severe exacerbations in the previous year

SECONDARY OUTCOMES:
Evolution of the number of severe exacerbations, defined as use of systemic corticosteroids during at least 3 days or hospitalizations or emergency visits due to asthma with use of systemic corticosteroids | Every 3 months during the study (up to 15 months)
Evolution of the frequency of self-reported adverse event of inhaled therapy for asthma | Every 3 months during the study (up to 15 months)
Evolution of treatment compliance measured by the Mediation Adherence Report Scale (MARS) and by pharmacy records | Every 3 months during the study (up to 15 months)
Evolution of the asthma control measured by the Asthma Control Questionnaire (ACQ) | Every 3 months during the study (up to 15 months)
Evolution of the asthma control measured by the Asthma Control Test (ACT) | Every 3 months during the study (up to 15 months)
Evolution of the asthma related quality of life by the mini-Asthma Quality of Life Questionnaire (miniAQLQ) | Every 3 months during the study (up to 15 months)
Evolution of the Fractional Exhaled Nitric Oxide (FeNO) | Every 3 months during the study (up to 15 months)
Evolution of lung function measured by percentage of predicted Forced Expiratory Volume in 1 second (%FEV1) | Every 3 months during the study (up to 15 months)
Evolution of lung function measured by Forced Expiratory Volume in 1 second (FEV1) divided by Forced Vital Capacity (FVC) | Every 3 months during the study (up to 15 months)
Evolution of lung function measured by reversibility to Short Acting Beta2-Agonists (SABA) | Every 3 months during the study (up to 15 months)
Evolution of inflammatory blood markers : blood cell count, fibrinogen, C-Reactive Protein (CRP) | Every 3 months during the study (up to 15 months)
Evolution of sputum markers of inflammation : rates of neutrophils, eosinophils, macrophages, lymphocytes, epithelial cells | Every 3 months during the study (up to 15 months)
Evolution of the number of moderate exacerbations, defined as the number of visits to an emergency room, the number of unscheduled doctor or pneumologist visits, and increases in reliever use | Every 3 months during the study (up to 15 months)
Evolution of the score of ICQ-S ("Inhaled Corticosteroids side-effect Questionnaire") | Every 3 months during the study (up to 15 months)
Check of the inhalation technique | Every 3 months during the study (up to 15 months)

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Louis, MD-PhD, Principal Investigator — University of Liege
Locations (1):
- University Hospital of Liege, Liège, Belgium

REFERENCES:
- [Derived] Demarche S, Schleich F, Henket M, Paulus V, Louis R, Van Hees T. Step-down of inhaled corticosteroids in non-eosinophilic asthma: A prospective trial in real life. Clin Exp Allergy. 2018 May;48(5):525-535. doi: 10.1111/cea.13106. Epub 2018 Mar 6. PMID 29383782